CLINICAL TRIAL: NCT02170207
Title: Lansoprazole Intravenous 30 mg Specified Drug-use Survey [Acute Stress Ulcer and Acute Gastric Mucosal Lesions]
Brief Title: Takepron Intravenous 30 mg Specified Drug-use Survey [Acute Stress Ulcer and Acute Gastric Mucosal Lesions]
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 254-012; JapicCTI-142542 (Registry Identifier: JapicCTI); JapicCTI-R160830 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Acute Stress Ulcer and Acute Gastric Mucosal Lesions
Keywords: Pharmacological therapy
MeSH Terms: interventions — Lansoprazole; Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 30 mg of lansoprazole: 30 mg of lansoprazole is mixed in physiological saline (JP) or 5% glucose solution for injection (JP) and administered twice daily by drip infusion or dissolved in 20 mL of physiological saline (JP) or 5% glucose solution for injection (JP) and administered twice daily by direct slow intravenous injection.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — Lansoprazole 30 mg injection
  Other Names: Takepron 30 mg Injection

SUMMARY:
The purpose of this survey is to evaluate the safety (that is, frequency of adverse events) and efficacy (that is, hemostatic effect, rate of rebleeding after confirmation of hemostasis) of administration of lansoprazole intravenous 30 milligram (mg) (Takepron Intravenous 30 mg ) to a large number of participants with acute stress ulcer or acute gastric mucosal lesion in daily medical practice.

DETAILED DESCRIPTION:
This survey was designed to evaluate the safety (that is, frequency of adverse events) and efficacy (i.e., hemostatic effect, rate of rebleeding after confirmation of hemostasis) of administration of lansoprazole intravenous 30 mg (Takepron Intravenous 30 mg) to a large number of participants with acute stress ulcer or acute gastric mucosal lesion in daily medical practice.

For adults, 30 mg of lansoprazole is typically mixed in physiological saline (JP) or 5 percent (%) glucose solution for injection (JP) and administered twice daily by drip infusion or dissolved in 20 mL of physiological saline (JP) or 5% glucose solution for injection (JP) and administered twice daily by direct slow intravenous injection.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Participants with the following diseases for whom oral administration is not feasible:

Acute stress ulcer, and acute gastric mucosal lesions (both of which should be accompanied by bleeding).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute stress ulcer and acute gastric mucosal lesions
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative site in Japan from 29 January 2007 to 31 March 2010.
Pre-assignment Details: Participants with a historical diagnosis of acute stress ulcer or acute gastric mucosal lesion accompanied with bleeding, for whom oral administration of drug was not feasible were observed in a single treatment group to receive lansoprazole 30 milligrams (mg).
Groups:
- Lansoprazole: Lansoprazole 30 milligram (mg), injection or drip infusion, intravenous, twice daily for up to 7 days followed by an observation period after the end of treatment for 8 weeks .
Period: Overall Study
Arm/Group | Lansoprazole
Started | 63
Completed | 58
Not Completed | 5
Not completed — Case report forms unavailable | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Arm/Group | Lansoprazole
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (16.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 36
Pregnancy Status [Number; unit: participants] — This baseline characteristic was analyzed only in female participants.
  participants
    Not pregnant | 22
    Pregnant | 0
Target Disease [Number; unit: participants] — This baseline characteristic was analyzed for participants who were suffering from disease being targeted in the study, which were acute stress-induced ulcer and acute gastric mucosal lesion.
  participants
    Acute Stress-Induced Ulcer | 46
    Acute Gastric Mucosal Lesion | 12
Healthcare Category [Number; unit: participants] — Participants were categorized as outpatient and inpatient. This baseline characteristic was analyzed for inpatient participants.
  participants | 58
Predisposition to Hypersensitivity [Number; unit: participants] — This baseline measure was analyzed in participants who had a tendency of suffering from hypersensitivity.
  participants
    No | 54
    Yes | 4
Helicobacter Pylori Infection [Number; unit: participants] — This baseline characteristic was analyzed in participants who tested either positive (had infection) or negative (did not have infection) for helicobacter pylori infection.
  participants
    Positive | 20
    Negative | 16
    Unknown | 22
Alcohol consumption [Number; unit: participants]
  Alcohol Consumer | 15
  Alcohol Non-Consumer | 38
  Unknown | 5
Smoking [Number; unit: participants]
  Smoker | 14
  Non-Smoker | 40
  Unknown | 4
Medical History [Number; unit: participants]
  Had medical history | 30
  Did not have medical history | 28
Breakdown of Medical History [Number; unit: participants] — This baseline characteristic was analyzed in participants who had a medical history of peptic ulcer or upper gastrointestinal bleeding or cerebrovascular accident or malignant tumor or hepatic dysfunction or renal dysfunction or diabetes mellitus or cardiac disorders or hypertension or any other type of disease. Participants may be represented in more than 1 category.
  participants
    Peptic ulcer | 13
    Upper gastrointestinal bleeding | 1
    Cerebrovascular accident | 4
    Malignant tumor | 3
    Hepatic dysfunction | 3
    Renal dysfunction | 0
    Diabetes mellitus | 2
    Cardiac disorders | 2
    Hypertension | 0
    Other | 11
Medical Complications [Number; unit: participants]
  Had Complications | 28
  Had no Complications | 30
Breakdown of Complications [Number; unit: participants] — This baseline characteristic was analyzed in participants who had hypertension, cardiac disorders, diabetes mellitus, hepatic dysfunction, anemia, malignant tumor, cerebrovascular accident, renal dysfunction and any other medical complications. Participants may be represented in more than 1 category.
  participants
    Hypertension | 8
    Cardiac disorders | 4
    Diabetes mellitus | 5
    Hepatic dysfunction | 3
    Anemia | 4
    Malignant tumor | 2
    Cerebrovascular accident | 1
    Renal dysfunction | 1
    Other | 18
Emotional Stress [Number; unit: participants]
  Had Stress | 29
  Had no Stress | 29
Breakdown of Drugs [Number; unit: participants] — The baseline characteristic was analyzed in participants who consumed non steroidal anti-inflammatory drugs, platelet aggregation inhibitors, anticoagulants, and steroids that affected the coagulation system during the month prior to administration of study drug. Participants may be represented in more than 1 category.
  participants
    Non Steroidal Anti-Inflammatory Drugs | 7
    Platelet aggregation inhibitors | 5
    Anticoagulants | 3
    Steroids | 0
    Other | 1
Prior Consumption of Drugs Affecting Coagulation System [Number; unit: participants] — The baseline characteristic was analyzed in participants who consumed drugs that affected the coagulation system during the month prior to administration of study drug.
  participants
    Had consumption | 12
    Had no consumption | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AEs) which are in the investigator's opinion of causal relationship to the study treatment. AEs are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to Week 9
Population: The safety analysis set was defined as all participants who were enrolled and completed the study.
Measure: Number; unit: participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 58
participants | 0

2. Secondary Outcome: Percentage of Participants With Observed Hemostatic Effect
Description: Hemostatic effect was categorized on the basis of degree of improvement as: markedly improved, moderately improved, slightly improved and poor in the participants with observed hemostatic effect. Efficacy rate was reported as percentage of participants showing efficacy and was calculated as the sum of percentage of number of participants reporting markedly improved + moderately improved + slightly improved divided by the percentage of total number of participants with observed hemostatic effect.
Time Frame: Baseline up to Week 9
Population: The efficacy assessment population was defined as participants who completed the study and had efficacy data at baseline and post-baseline time points available.
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 58
percentage of participants | 96.6

3. Secondary Outcome: Percentage of Participants With Confirmed Hemostatic Effect
Description: Hemostatic effect was categorized on the basis of degree of improvement as: markedly improved, moderately improved, slightly improved and poor in the participants with confirmed hemostatic effect by endoscopy. Efficacy rate was reported as percentage of participants showing efficacy and was calculated as the sum of percentage of number of participants reporting markedly improved + moderately improved + slightly improved divided by the percentage of total number of participants with confirmed hemostatic effect.
Time Frame: Baseline up to Week 9
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 45
percentage of participants | 95.6

4. Secondary Outcome: Percentage of Participants With Confirmed Hemostatic Effect Who Experienced Rebleeding During Treatment
Description: Rebleeding rate was reported as percentage of participants who experienced rebleeding after confirmed hemostasis by endoscopy during treatment with lansoprazole. It was calculated by dividing the percentage of the number of participants who experienced rebleeding after hemostasis divided by the total number of participants with confirmed hemostasis.
Time Frame: Baseline up to Week 9
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 43
percentage of participants | 0

5. Secondary Outcome: Percentage of Participants With Confirmed Hemostatic Effect Who Experienced Rebleeding After the Completion of Treatment
Description: Rebleeding rate was reported as percentage of participants who experienced rebleeding after confirmed hemostasis by endoscopy and was calculated at 8 weeks after the completion of treatment with lansoprazole. It was calculated by dividing the percentage of the number of participants who experienced rebleeding after hemostasis divided by the total number of participants with confirmed hemostasis.
Time Frame: Week 17 (8 weeks after the last dose of study drug)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lansoprazole
Number analyzed (Participants) | 30
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 17
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in this study.
Arm/Group | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 0/58
Other Adverse Events (participants affected / at risk) | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.